CLINICAL TRIAL: NCT00000695
Title: Open Label Phase I Study To Evaluate the Safety of Combination Therapy With AZT and Interferon-Beta in Patients With AIDS Related Kaposi's Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 057; 11031 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Sarcoma, Kaposi; HIV Infections
Keywords: Drug Evaluation; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; Zidovudine; Interferon Type I
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Interferon beta-1b; Zidovudine

INTERVENTIONS:
Drug: Interferon beta-1b
Drug: Zidovudine

SUMMARY:
To determine the highest tolerated dose of the safety and tolerance of interferon beta (IFN-B) when it is given at the same time as zidovudine (AZT) to patients with early AIDS related Kaposi's sarcoma. In addition, the studies will determine preliminary data on response, immune function, and subcutaneous absorption.

IFN-B has demonstrated a dose-dependent ability to suppress the replication of HIV in the test tube. In addition, previous studies have shown AZT to be an effective inhibitor of HIV reverse transcriptase; Phase I and II study benefits of AZT treatment include increased objective clinical improvement, decreased mortality rate, and decreased incidence of opportunistic infections. Long-term AZT use, however, presents possible limitations secondary to intolerance. This study, therefore, will investigate the potential antiviral activities of a combination of IFN-B and AZT to determine the safety and efficacy of such treatment in patients with AIDS related Kaposi's sarcoma. It is believed that combination drug therapy consisting of low doses of each drug will reduce the potential of toxicity, treatment failures, and disease recurrences resulting from drug-resistant virus mutants.

DETAILED DESCRIPTION:
IFN-B has demonstrated a dose-dependent ability to suppress the replication of HIV in the test tube. In addition, previous studies have shown AZT to be an effective inhibitor of HIV reverse transcriptase; Phase I and II study benefits of AZT treatment include increased objective clinical improvement, decreased mortality rate, and decreased incidence of opportunistic infections. Long-term AZT use, however, presents possible limitations secondary to intolerance. This study, therefore, will investigate the potential antiviral activities of a combination of IFN-B and AZT to determine the safety and efficacy of such treatment in patients with AIDS related Kaposi's sarcoma. It is believed that combination drug therapy consisting of low doses of each drug will reduce the potential of toxicity, treatment failures, and disease recurrences resulting from drug-resistant virus mutants.

Patients undergo evaluations to determine the extent of their disease and the status of their immune system. Patients then receive IFN-B subcutaneously once a day at one of three different dose levels. Patients also take AZT at 1 of 2 doses. The first 12 patients are treated with the lower dose of AZT. The first 4 patients are entered at level 1 of IFN-B. If no dose-limiting toxicity is seen in these 4 patients after 2 weeks of therapy, 4 patients are then enrolled at level 2 of IFN-B. The study proceeds in this manner until the highest tolerated dose or level 3 is reached. If both drugs are tolerated, patients then remain on both medications as long as they continue to tolerate the medications and show some improvement in either antiviral response, immune response, or clinical response for as long as 24 weeks. The initial three doses of IFN-B are given to each patient at the study site during which time the patient is trained to self-administer the IFN-B. Patients are then seen weekly for 4 months and every 2 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria

Concurrent Treatment:

Allowed:

* Local radiotherapy or laser therapy to cosmetically apparent Kaposi's lesions, provided the dose to any one lesion does not exceed 3000 gray and the total surface area of all lesions treated does not exceed 10 cm2 during the course of the trial.

Patients must demonstrate the following clinical and laboratory findings:

* Positive for HIV by federally licensed ELISA test.
* Acceptable bone marrow function.
* Acceptable renal function.
* Acceptable hepatic function.

Exclusion Criteria

Concurrent Medication:

Excluded:

* Other potentially antiretroviral compounds.

Patients will be excluded from the study for the following reasons:

* Concurrent, active opportunistic infections requiring therapy.
* Extensive Kaposi's sarcoma with more than 100 cutaneous lesions, requiring systemic chemotherapy, prior treatment with more than one chemotherapy regimen, excluding intralesional therapy, or symptomatic visceral Kaposi's sarcoma.
* Evidence of clinically significant cardiac dysfunction (New York Heart Association grade III or IV).
* History of malignant neoplasms other than nonmelanomatous skin cancer or cancer in situ of the cervix.
* Proteinuria of 2+ or greater and/or 24-hour urine protein of greater than 1.

Prior Medication:

Excluded:

* More than one chemotherapy regimen for Kaposi's sarcoma.
* Any interferon preparation or zidovudine (AZT).
* Excluded within 30 days of study entry:
* Other immunomodifiers.
* Acyclovir.
* Other investigational drugs.
* Excluded within 60 days of study entry:
* Cytotoxic therapy.

Patients may not have any of the following diseases or symptoms:

* Development of an AIDS-defining opportunistic infection, other than oral thrush or localized zoster.
* Non-Kaposi's sarcoma, AIDS-defining malignancy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36
Dates: Study Completion 1991-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: S Miles, Study Chair
Locations (4):
- United States (4):
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - USC School of Medicine / Norris Cancer Hosp, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - Northwestern Univ Med School, Chicago, Illinois

REFERENCES:
- [Background] Stavermann T, Bauer G, Ruess A. Recombinant interferon-beta in the therapy of advanced AIDS-related Kaposi's sarcoma. Int Conf AIDS. 1993 Jun 6-11;9(1):402 (abstract no PO-B12-1600)
- [Background] Miles S, Levine A, Feldstein M, Carden J, Cabriallas S, Marcus S, Mitsuyasu R, Gill P. Open-label phase I study of combination therapy with zidovudine and interferon-beta in patients with AIDS-related Kaposi's sarcoma: AIDS Clinical Trials Group Protocol 057. Cytokines Cell Mol Ther. 1998 Mar;4(1):17-23. PMID 9557213